CLINICAL TRIAL: NCT04174066
Title: From Immune System Damage to Podocyte Cell Damage: Prospective Database and Biological Collection of Patients (Children and Adults) With Minimal Glomerular Injury Nephrotic Syndrome (MGLS) and Primary Segmental and Focal Hyalinosis (HSFP)
Brief Title: From Immune System Damage to Podocyte Cell Damage: Prospective Database and Biological Collection of Patients (Children and Adults) With MGLS and HSFP
Acronym: BiobankSNI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-PP-16
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-11

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: whole blood / plasma / serum collected specifically for the Biobank but during a blood test planned in the follow-up of patients.
  Tissue sample: slide of biopsies taken during the treatment Excreta: urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SNLGM: 70 patients with an SNLGM
  Interventions: Other: blood sample; Other: tissue sample; Other: excreta
- primary FSH: 74 with a primary FSH
  Interventions: Other: blood sample; Other: tissue sample; Other: excreta

INTERVENTIONS:
Other: blood sample — blood sample during planned in the follow-up of patients.
Other: tissue sample — tissue sample during planned in the follow-up of patients.
Other: excreta — urine sample during planned in the follow-up of patients.

SUMMARY:
Idiopathic Nephrotic Syndrome (INS) is a kidney disease characterized by massive proteinuria and hypoalbuminemia. It includes two anatomopathological entities: nephrotic syndrome with minimal glomerular lesions (SNLGM) and primary segmental and focal hyalinosis (PHF). Renal biopsy reveals a fusion of the feet of the podocytes without inflammatory lesions or deposits of immune complexes. Clinical and experimental observations strongly suggest that the immune system and podocyte dysfunction are the two facets of the disease. There are currently no clinical or biological markers to predict the diagnosis of corticosteroid sensitivity, corticosteroid dependence, or risk of recurrence of kidney disease after kidney transplantation. To our knowledge, no prospective studies have been designed to study both immune system alterations and podocyte damage as well as genetic predisposition variants in NIS. Therefore, the use of steroids/immunosuppressive agents is purely empirical with a multitude of side effects.

The objective is to identify and test new therapeutic targets rather than conducting new trials with existing treatments, using either drug candidates or molecules selected by high throughput screening of libraries of repositioning molecules using an appropriate read-out. The biobank may also be used to analyze the effects of conventional treatments on identified new biomarkers. We expect the project to produce original and patentable results with subsequent valuation. Patentability will be anticipated before any publication on the subject. The patent and valorization cells of hospitals, INSERM and Universities will be involved in the results as soon as they are obtained.

ELIGIBILITY:
Inclusion Criteria:

* First episode of idiopathic nephrotic syndrome in a child aged 12 months to 18 years with a weight > 10 kg and biologically defined as proteinuria > 0.20 g / mmol creatinuria and hypoalbuminemia <25 g / mmol
* First episode of NIS defined in adults as albumin level <30 g / L and a urinary protein/creatinine ratio (UPCR) ≥ 300 mg / mmol systematically associated with the performance of a renal anatomopathological examination and characterized by the absence of identifiable lesions by light microscopy (SNLGM) or the presence of HSF lesions.
* For adults: signed informed consent to participate in the study
* For children: patients will be informed and a written informed consent form will be signed by both parents of the children at inclusion
* Patients affiliated to the French health system

Exclusion Criteria:

* Patients who have previously received corticosteroids and/or immunosuppressants
* Patients with reduced CH50 and/or low C3 and/or low C4 and/or low C4 (in some cases increased sC5b9 and/or presence of a C3 nephritic Factor; an anti-C3b...)
* SNLGM resulting from a secondary process (lymphoid hematopathies or neoplasia) or occurring following the administration of a treatment known to be associated with an SNLGM (lithium, interferon, non-steroidal anti-inflammatory drugs)
* Non-primary FHH (absence of Nephrotic Syndrome, etiological assessment revealing FHH secondary to an identified cause (genetic or not), no introduction of corticosteroids or immunosuppressants as first-line treatment)
* Positive serological screening test for HIV, hepatitis B or C
* Positive immunological tests for antinuclear and anti-DNA antibodies or anti-PLA2R1 and anti-THSD7A
* Patient under guardianship or curatorship

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with Idiopathic Nephrotic Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
number of biological samples | 5 years
  establish in each centre a prospective collection of blood, urine and kidney biopsy samples sampled and stored in accordance with standard operating procedures, supported by a harmonized clinical and biological database

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nice Hospital, Nice
  - APHP, Paris

IPD SHARING:
Plan to Share IPD: No